CLINICAL TRIAL: NCT01276431
Title: Norspan Efficacy and Safety Among Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUP4504; 2010-020748-37 (EudraCT Number)
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthritis Pain of the Hip and or Knee

ARMS (1):
- Buprenorphine transdermal patch (Other): For two age groups: 50-60 years and >= 75 years of age
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch

SUMMARY:
An open label, multi-centre, prospective age-group-controlled study to evaluate efficacy and safety of buprenorphine transdermal patches in subjects with chronic, moderate to severe osteoarthritis pain of the hip and/or knee.

ELIGIBILITY:
Summary Criteria for Inclusion:

1. Males and females aged 50-60 or ≥ 75 years.
2. Subjects with clinical diagnosis of osteoarthritis in knee and/or hip including fulfilment of ACR-criteria and radiographic evidence not older than one year.
3. Subjects with a moderate to severe pain, confirmed by a BS-11 score ≥ 4 for their pain on average during the last seven days of the Screening Phase in their primary OA-site at the Baseline Visit.

Summary Criteria for Exclusion:

1. Subjects recording < 4 on average during the Screening Phase on the BS-11 scale.
2. Subjects treated with high-potent opioid analgesics (e.g. morphine, fentanyl, oxycodone, methadone, hydromorphone, ketobemidone, buprenorphine) for their osteoarthritis pain.
3. Subjects treated with a regular dose for > 1 week of tramadol, codeine or dextropropoxyphene within 1 month before screening visit.
4. Subjects who require NSAID treatment (except aspirin for cardiovascular indications) or cox-2-inhibitors during the study period.
5. Subjects with history of, or ongoing, chronic condition(s), in addition to osteoarthritis, requiring frequent analgesic therapy (e.g. frequent headaches, frequent migraine, gout, rheumatoid arthritis).
6. Subjects scheduled for surgery that would fall within the study period.
7. Subjects who currently abused substance or alcohol, or subjects who, in the opinion of the Investigator, have demonstrated addictive or substance abuse behaviours.
8. Subjects with cancer (except basal cell carcinoma) or history of cancer in the last 5 years (except treated basal cell carcinoma).
9. Untreated depression or other psychiatric disorder in such way that participation in the study may, in the opinion of the Investigator, pose an unacceptable risk to the subject.
10. Subjects who are currently taking hypnotics, anxiolytics or other central nervous system depressants that, in the Investigator's opinion, may pose a risk of additional CNS depression with study medication.
11. Subjects who are currently taking adjuvant analgesics such as antidepressants and anti-convulsants.
12. Dermatological disorder or non-intact skin at any relevant patch application site that precludes proper placement and/or rotation of patch placement.
13. Subjects who had received an intra-articular steroid injection within 6 weeks prior Screening Visit or subjects who require steroid treatment (oral, intra-muscular, intra-venous, intra-articular, epidural or other corticosteroid injections) during the study period.
14. Subjects with joint evacuation 6 weeks prior Screening Visit and during the study.
15. Subjects who are currently taking monoamine oxidase inhibitors (MAOI's) or have taken MAOI's within 2 weeks before Screening Visit.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Box Scale-11 (BS-11) pain scores (pain on average during the last seven days, mean change from Baseline to Completion (fulfilled all visits in the study).

SECONDARY OUTCOMES:
Western Ontario & McMaster Universities OA Index
European QOL Health Questionnaire
Sleep disturbance & quality of sleep questions
Patients global assessment of pain relief
Investigators global assessment of pain relief
Incidence of rescue medication

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Professor Jon Karlsson, Mölndal
  - Dr Bengt Olav Tengmark, Stockholm

REFERENCES:
- [Background] Karlsson J, Soderstrom A, Augustini BG, Berggren AC. Is buprenorphine transdermal patch equally safe and effective in younger and elderly patients with osteoarthritis-related pain? Results of an age-group controlled study. Curr Med Res Opin. 2014 Apr;30(4):575-87. doi: 10.1185/03007995.2013.873714. Epub 2013 Dec 23. PMID 24320787